CLINICAL TRIAL: NCT03041363
Title: Treatment Development of Triheptanoin (C7) for Glucose Transporter Type I Deficiency (G1D): A Phase I Maximum Tolerable Dose Trial
Brief Title: Treatment Development of Triheptanoin (G1D)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juan Pascual (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Juan Pascual, PROFESSOR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 062016-105; R01NS094257 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy; GLUT1DS1; Glut1 Deficiency Syndrome 1, Autosomal Recessive; Glucose Metabolism Disorders; Glucose Transport Defect; Glucose Transporter Type 1 Deficiency Syndrome; Glucose Transporter Protein Type 1 Deficiency Syndrome
MeSH Terms: conditions — Epilepsy; Glucose Metabolism Disorders; Glycogen Storage Disease Id; Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: The trial will use an open-label, standard 3+3 phase 1 design for determining the MTD of orally administered C7 in G1D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Triheptanoin (Experimental): Dose 1 C7 administered as 40% daily caloric intake. Dose 2. C7 administered as 45% daily caloric intake.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin will be administered for 7 days 4 times daily.
  Other Names: C7

SUMMARY:
To determine the maximum tolerated dose (MTD), as a percentage of calories consumed, of triheptanoin (C7 oil; C7) in a pediatric and adult patient population genetically diagnosed with glucose transporter type 1 deficiency disorder (G1D).

DETAILED DESCRIPTION:
The trial will use an open-label, standard 3+3 phase I design for determining the MTD of orally-administered C7 in G1D.

Triheptanoin: a triglyceride oil containing three odd-carbon chain-length fatty acids (i.e., a triglyceride of 7-carbon heptanoic acid). Triheptanoin will be taken 4 times per day (approximately every 6 hours) by mouth. it is dosed 4 times per day, divided evenly, and the total C7 daily dose will re-place 40% or 45% (depending on group) of the daily caloric intake from fat in the usual diet, based on current protocol guidelines. The oil should be taken approximately one hour before meals, and will be mixed with fat-free, sugar-free yogurt or pudding for administration.

Up to thirty-six subjects will be enrolled in a 10-day maximum tolerable dose trial of C7. Initiation of C7 dosing will be conducted in the Children's Medical Center Dallas ambulatory Care Pavilion neurology Clinic. Subjects will be provided with C7 oil to take over the 7 days of administration.

Subjects will not be required to stop other medications. Subjects will be directed to maintain their usual medications, including rescue seizure medications, as necessary for the course of the study. Subjects may have any clinical medical records transferred back to their referring physician at completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glucose transporter type I deficiency (G1D) confirmed by genotyping or PET scan of the brain.
* Stable on no dietary therapy other than Modified Atkins diet (i.e., on no dietary therapy for 1 month, including, but not limited to, medium chain triglyceride therapy).
* Males and females 2 years 6 months to 35 years 11 months old, inclusive.

Exclusion Criteria:

* Subjects with a history of life-threatening seizure episodes, including but not limited to status epilepticus and cardiac arrest.
* Subjects with evidence of independent, unrelated metabolic and/or genetic disease.
* Subjects with a body mass index (BMI) greater than or equal to 30.
* Subjects with a chronic gastrointestinal disorder, such as irritable bowel syndrome, Crohn's disease, or colitis, which could increase the subject's risk of developing diarrhea or stomach pain.
* Subjects currently on dietary therapy (i.e., ketogenic diet, medium chain triglyceride-supplemented diets, Atkins diet, low glycemic index diet, and related diets).
* Women who are pregnant or breast-feeding may not participate.
* Women who plan to become pregnant during the course of the study, or who are unwilling to use birth control to prevent pregnancy (including abstinence) may not participate.
* Females age 10 and over will be asked to provide a urine sample for a pregnancy test via dipstick.
* Subjects will be asked to agree to abstinence or another form of birth control for the duration of the study.
* Allergy/sensitivity to C7.
* Previous treatment with C7 one month prior to enrollment.
* Treatment with medium chain triglycerides in the last 30 days.
* Subjects exhibiting signs of dementia, or diagnosed with any degenerative brain disorder (such as Alzheimer's disease) that would confound assessment of cognitive changes, in the opinion of the investigator.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of 1 parent or legal guardian/representative to give written informed consent.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose trial | medication taken daily for 7 days.
  To determine the MTD as a percentage of calories consumed in pediatric and adult patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pascual, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascual JM, Liu P, Mao D, Kelly DI, Hernandez A, Sheng M, Good LB, Ma Q, Marin-Valencia I, Zhang X, Park JY, Hynan LS, Stavinoha P, Roe CR, Lu H. Triheptanoin for glucose transporter type I deficiency (G1D): modulation of human ictogenesis, cerebral metabolic rate, and cognitive indices by a food supplement. JAMA Neurol. 2014 Oct;71(10):1255-65. doi: 10.1001/jamaneurol.2014.1584. PMID 25110966
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Pascual JM, Ronen GM. Glucose Transporter Type I Deficiency (G1D) at 25 (1990-2015): Presumptions, Facts, and the Lives of Persons With This Rare Disease. Pediatr Neurol. 2015 Nov;53(5):379-93. doi: 10.1016/j.pediatrneurol.2015.08.001. Epub 2015 Aug 10. PMID 26341673
- [Derived] Malaga I, Avila A, Primeaux S, Kallem RR, Roe CR, Putnam WC, Park JY, Shinnar S, Ahn C, Pascual JM. Maximum dose, safety, tolerability and ketonemia after triheptanoin in glucose transporter type 1 deficiency (G1D). Sci Rep. 2023 Mar 1;13(1):3465. doi: 10.1038/s41598-023-30578-z. PMID 36859467